CLINICAL TRIAL: NCT06263127
Title: The Effectiveness of Prefeeding Oral Stimulation and Infant Massage on Preterm Infants in the Neonatal Care Unit
Brief Title: Sensory Motor Interventions on Preterm Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH112-REC2-104
Record Dates: First submitted 2024-01-10; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Preterm Infants
Keywords: NICU; Massage; Preterm infants; oral stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OS group (Experimental): The participants receive the prefeeding oral stimulation intervention twice a day,10 days.
  Interventions: Behavioral: oral stimulation
- OS+ IM group (Experimental): The participants receive both prefeeding oral stimulation and infant massage once a day, in random order, 10 days.
  Interventions: Behavioral: oral stimulation; Behavioral: infants massage

INTERVENTIONS:
Behavioral: oral stimulation — Prefeeding OS is a 5-minute oral sensorimotor intervention, containing peri- and intra-oral stimulation for 3 minutes and pacifier sucking for 2 minutes.
  Other Names: oral sensoriomotor stimulation
Behavioral: infants massage — IM is a 15-minute intervention, involving 5-min manual stroking on the infant's head, neck, back, upper limbs, and lower limbs twice and 5-min gentle flexion and extension exercises on the infant's arms and legs.
  Other Names: body massage
  Arms: OS+ IM group

SUMMARY:
Preterm infants experiencing bottle feeding difficulties will be included in this study. Two distinct interventions, oral stimulation (OS) and infant massage (IM), will be administered in this study. The objective of this clinical trial is to compare the effectiveness of these two approaches, either individually or in combination, in improving the feeding performance and development of participants.

DETAILED DESCRIPTION:
Currently, two rehabilitation approaches, Prefeeding oral stimulation (OS) and infant massage (IM), are often used by health professionals to facilitate preterm infants' oral feeding abilities. The purpose of this study is to compare the effectiveness of prefeeding OS and the combined approach of prefeeding OS and IM in improving feeding performance and development of preterm infants. Participants will randomly allocated to two groups and receive either OS or combined OS plus IM. Prefeeding OS is a 5-minute oral sensorimotor intervention, containing peri- and intra-oral stimulation for 3 minutes and pacifier sucking for 2 minutes. IM is a 15-minute intervention, including 5-min manual massage on the infant's head, neck, back, upper limbs, and lower limbs twice and 5-min passive exercise of moving the infant's arms and legs once. The OS group will receive OS twice a day for 10 days. The combined group will receive OS once and IM once a day for 10 days.

Both groups will undergo a bottle feeding assessment before, mid-term, and after the intervention period. Neurodevelopmental assessments will be conducted before and after the intervention period. Additionally, the investigator will conduct chart review to collect participants' birth and medical data. The primary outcomes are feeding performance parameters (e.g., the rate of milk transfer in the first 5 minutes of feeding, total oral intake volume, and milk leakage during bottle feeding) and neurodevelopment outcomes. Secondary outcomes include weight gain and hospital stay. Furthermore, a follow-up evaluation on feeding questionnaire at home and sensory processing function will be conducted when the infants reach three months of corrected age.

ELIGIBILITY:
Inclusion Criteria:

1. < 34 weeks' gestational age
2. 34~40 weeks' postmenstrual age at enrollment
3. being fed by oral for at least 2 days but with poor feeding performance defined as consuming less than 80% of the prescribed volume for the half or more feedings
4. weaning the ventilator and maintaining stable physiological status

Exclusion Criteria:

1. Congenital anomalies
2. Confirmed or suspected chromosomal or genetic abnormalities
3. Unsolved seizure, sepsis, necrotizing enterocolitis(NEC)

Max Age: 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Oral intake | the 1st, 8th, and 14th day of the intervention period
  The volume of oral intake in the feeding
Transition time of oral feeding | from the date of the first day of the intervention until the date of full oral feeding, assesed up to 4 weeks
  the number of days from the first day of the intervention to the day at full oral feeding

SECONDARY OUTCOMES:
weight gain | 14 days
  weight gain from the first day to the last day of the intervention period
Hospital stay | from the date of the first day of the intervention until the date of hospital discharge, assessed up to 6 weeks
  the number of days from the first day of the intervention to the day of discharge
Neonatal Neurobehavioral Examination-Chinese Version(NNE-C) | the 1st and 14th day of the intervention period
  It consists of three subtests: (1) Muscle Tone and Movement Patterns (12-36 points), (2) Primitive Reflexes (13-39 points), and (3) Behavioral Responses (12-36 points). A higher score means more mature motor pattern.
Infant/Toddler Sensory Profile-Chinese Version(ITSP-C) | conducted at around 3 months of corrected age
  A self-reported questionnaire completed by the primary caregiver will be used to assess sensory processing of infants from birth to three years old. It consists of 5 subscales: General Perception, Auditory Processing, Visual Processing, Tactile Processing, and Vestibular Processing. The items of the five subscales can be classified into 4 quadrants: Low registration (13-65 points), sensory seeking (6-30 points), sensation sensitivity (12-60 points), and sensory avoiding (5-25 points). A lower score means a stronger sensory quadrant pattern.
Premature Bottle Feeding Questionnaire(PBFQ) | conducted at around 3 months old of corrected age
  A self-reported questionnaire consists of 15-item feeding problematic behaviors. The primary caregiver will fill out each question using a 4-point scale according to the infant's feeding performance at home. The feeding score is from 15 to 60 points. A higher score means poorer feeding performance.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No